CLINICAL TRIAL: NCT02640664
Title: RAINBOW Extension Study: an Extension Study to Evaluate the Long Term Efficacy and Safety of RAnibizumab Compared With Laser Therapy for the Treatment of INfants BOrn Prematurely With Retinopathy of Prematurity
Brief Title: Rainbow Extension Study
Acronym: RainbowExt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002H2301E1; 2014-004048-36 (EudraCT Number)
Record Dates: First submitted 2015-12-01; First posted 2015-12-29 (Estimated); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: open-label,; long-term,; extension study,; intravitreal ranibizumab,; laser ablation therapy,; retinopathy of prematurity,; preterm infants,; RAINBOW
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ranibizumab 0.2 mg (Experimental): 1 intravitreal injection in both eyes on Day 1 (Baseline), with up to 2 re-treatments allowed for each eye if required
  Interventions: Drug: Ranibizumab
- Ranibizumab 0.1 mg (Experimental): 1 intravitreal injection in both eyes on Day 1 (Baseline), with up to 2 re-treatments allowed for each eye if required
  Interventions: Drug: Ranibizumab
- Laser therapy (No Intervention): Laser therapy

INTERVENTIONS:
Drug: Ranibizumab — 1 intravitreal injection in both eyes on Day 1 (Baseline), with up to 2 re-treatments allowed for each eye if required
  Arms: Ranibizumab 0.1 mg; Ranibizumab 0.2 mg

SUMMARY:
The purpose of this study was to evaluate the long term efficacy and safety of intravitreal ranibizumab compared with laser ablation therapy in patients who were treated for retinopathy of prematurity (ROP) in the core study CRFB002H2301 (NCT02375971)

DETAILED DESCRIPTION:
This was a multicenter, open-label extension study where the Visual Acuity (VA) assessment at the child's 5th birthday visit was performed. The study had 2 distinct periods (Epochs). Treatment with study ranibizumab (either as retreatment after ranibizumab had already been injected in the same eye or as switch ranibizumab treatment from study laser therapy administered in the core study) was permitted for eligible eyes with recurrence/worsening of ROP up to and including Week 40 from the baseline visit in the core study (Epoch 1). The remainder of the extension study up to the 5th birthday visit (Epoch 2) was observational, with no study treatment planned to be administered.

In the core study, patients were randomized to 1 of the 3 treatment arms (ranibizumab 0.2 mg, ranibizumab 0.1 mg, and laser). Treatment arm assignment and patient identifier in the extension study remained the same as in the core study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s), in compliance with local requirements
* The patient successfully completed the core study H2301, as defined by providing assessments at the Visit 112 (the last scheduled visit in the core study) or, if appropriate, at the last of the additional assessment visits as per protocol in H2301, whichever was latest
* The patient received study treatment in both eyes at baseline of study H2301

Exclusion Criteria:

* Patient had a medical condition or personal circumstance which precluded study participation or compliance with study procedures, as assessed by the Investigator
* Patient had been discontinued from the core study H2301 at any time

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (71):
- United States (9):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Morgantown, West Virginia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Zagreb, Croatia
- Czechia (3):
  - Novartis Investigative Site, Praha 4 - Podoli, Czech Republic
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Koebenhavn Ø, Denmark
- Novartis Investigative Site, Alexandria, Egypt
- Novartis Investigative Site, Tallinn, Estonia
- France (2):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Marseille
- Novartis Investigative Site, Hanover, Germany
- Greece (3):
  - Novartis Investigative Site, Ampelokipoi, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- India (6):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Vanchiyoor, Thiruvanantapuram
  - Novartis Investigative Site, New Delhi
- Italy (4):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Fiumicino, RM
  - Novartis Investigative Site, Roma, RM
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Yachiyo, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Zentsujichó, Kagawa-ken
  - Novartis Investigative Site, Shimajiri-Gun, Okinawa
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Sumida-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Novartis Investigative Site, Kaunas, LTU, Lithuania
- Malaysia (2):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, Kota Kinabalu, Sabah
- Romania (3):
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Russia (4):
  - Novartis Investigative Site, Cheboksary
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Bratislava, Slovakia
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, Bakirkoy
  - Novartis Investigative Site, Meselik, Eskişehir
  - Novartis Investigative Site, Soguksu / Antalya, Turkey
- United Kingdom (2):
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Marlow N, Reynolds JD, Lepore D, Fielder AR, Stahl A, Hao H, Weisberger A, Lodha A, Fleck BW. Ranibizumab versus laser therapy for the treatment of very low birthweight infants with retinopathy of prematurity (RAINBOW): five-year outcomes of a randomised trial. EClinicalMedicine. 2024 Apr 11;71:102567. doi: 10.1016/j.eclinm.2024.102567. eCollection 2024 May. PMID 38638400
- [Derived] Marlow N, Stahl A, Lepore D, Fielder A, Reynolds JD, Zhu Q, Weisberger A, Stiehl DP, Fleck B; RAINBOW investigators group. 2-year outcomes of ranibizumab versus laser therapy for the treatment of very low birthweight infants with retinopathy of prematurity (RAINBOW extension study): prospective follow-up of an open label, randomised controlled trial. Lancet Child Adolesc Health. 2021 Oct;5(10):698-707. doi: 10.1016/S2352-4642(21)00195-4. Epub 2021 Aug 13. PMID 34391532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was carried out in Austria (2), Belgium (2), Croatia (1), Czech Republic (3), Denmark (1), Egypt (1), Estonia (1), France (2), Germany (1), Greece (3), Hungary (2), India (6), Italy (4), Japan (16), Lithuania (1), Malaysia (2), Romania (3), Russian Federation (5), Saudi Arabia (1), Slovakia (1), Taiwan (2), Turkey (3), United Kingdom (2), United States of America (9)
Pre-assignment Details: This study was not randomized. During Epoch 1 (starting at the baseline visit for the extension study up to 40 weeks from the baseline visit in the core study) participants continued to receive treatment as in the core study (NCT02375971). During Epoch 2 (starting at the end of Epoch 1 up to participant's 5th birthday) participants no longer received treatment (the study was observational)
Groups:
- Laser Therapy: Laser treatment to each eye on Day 1 (Baseline), with supplementary treatments allowed
Period: Epoch 1
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Started | 61 | 65 | 54
Completed (Number of subjects who completed post-treatment follow-up 1 (Epoch 1)) | 60 | 65 | 53
Not Completed | 1 | 0 | 1
Not completed — Withdrawal of informed consent | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1
Period: Epoch 2
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Started | 60 | 65 | 53
Completed (Number of subjects who completed post-treatment follow-up 2) | 54 | 55 | 47
Not Completed | 6 | 10 | 6
Not completed — Withdrawal of informed consent | 3 | 4 | 2
Not completed — Subject/guardian decision | 0 | 2 | 2
Not completed — Lost to Follow-up | 3 | 4 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy | Total
Number analyzed (Participants) | 61 | 65 | 54 | 180
Age, Continuous [Mean (Standard Deviation); unit: Weeks] — Age at extension baseline visit
  Weeks | 38.88 (7.316) | 40.16 (9.836) | 37.48 (8.745) | 38.92 (8.739)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 27 | 94
  Male | 29 | 30 | 27 | 86
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 38 | 40 | 32 | 110
  Black | 0 | 4 | 2 | 6
  Asian | 22 | 18 | 18 | 58
  Native American | 0 | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0
  Other | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA) of the Better-seeing Eye at the Participant's Fifth Birthday Visit - Comparison Between Treatment Arms
Description: The VA assessment at the child's 5th birthday visit was performed using Early Treatment Diabetic Retinopathy Study (ETDRS) methodology. VA measurements were taken in a sitting position at an initial test distance of 3 meters using Lea Symbols charts. Scores represented the number of optotypes (Lea symbols) the participant identified and ranged from 0 to 100, with higher scores indicating better visual acuity. VA was tested in each eye, using the child's current refractive index. The better-seeing eye was defined as the eye with the higher ETDRS score at the 5th birthday visit. If both eyes had the same ETDRS score, then the right eye was assigned as the better-seeing eye.
Time Frame: at the participant's fifth birthday visit (maximum 5 years and 4 months post core baseline visit)
Population: Extension Safety Set: defined as the subset of the participants from the Safety Set of the core study who entered the extension study and comprised data from both core and extension studies. The outcome measure included number of participants contributing to analysis.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 45 | 43 | 36
Score on a scale | 66.8 (1.95) | 64.6 (2.00) | 62.1 (2.18)
Statistical Analysis 1: Comparison: Ranibizumab 0.2 mg vs Laser Therapy; Test type: Superiority; ANOVA — primary endpoint in the extension study does not have p-values. It's a descriptive analysis; Mean Difference (Net) = 4.7, 95% CI 2-sided [-1.1 to 10.5], Standard Error of Mean 2.93
Statistical Analysis 2: Comparison: Ranibizumab 0.1 mg vs Laser Therapy; Test type: Superiority; ANOVA — primary endpoint in the extension study does not have p-values. It's a descriptive analysis; Mean Difference (Net) = 2.5, 95% CI 2-sided [-3.4 to 8.3], Standard Error of Mean 2.96
Statistical Analysis 3: Comparison: Ranibizumab 0.2 mg vs Ranibizumab 0.1 mg; Test type: Superiority; ANOVA — primary endpoint in the extension study does not have p-values. It's a descriptive analysis; Mean Difference (Net) = 2.2, 95% CI 2-sided [-3.3 to 7.8], Standard Error of Mean 2.79

2. Secondary Outcome: Number of Participants With Ocular Adverse Events (AEs) Regardless of Study Treatment or Procedure Relationship by Preferred Term
Description: Number of participants with ocular AEs starting during the core study and ongoing at extension baseline, or starting on/after extension baseline were reported.
Time Frame: throughout the study, approximately 5 years
Population: Extension Safety Set: defined as the subset of the patients from the Safety Set of the core study who entered the extension study and comprised data from both core and extension studies. The outcome measure included number of participants contributing to analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants | 19 | 26 | 22

3. Secondary Outcome: Number of Participants With Non-ocular Adverse Events (AEs) Regardless of Study Treatment or Procedure Relationship (Greater Than or Equal to 3% in Any Arm) by Preferred Term
Description: Number of participants with non-ocular adverse events regardless of study treatment or procedure relationship (greater than or equal to 3% in any arm) by preferred term were reported.
Time Frame: throughout the study, approximately 5 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants | 46 | 53 | 46

4. Secondary Outcome: Visual Acuity (VA) of the Worse-seeing Eye at the Participant's Fifth Birthday Visit - Comparison Between Treatment Arms
Description: The VA assessment at the child's 5th birthday visit was performed using Early Treatment Diabetic Retinopathy Study (ETDRS) methodology. VA measurements were taken in a sitting position at an initial test distance of 3 meters using Lea Symbols charts. Scores represented the number of optotypes (Lea symbols) the participant identified and ranged from 0 to 100, with higher scores indicating better visual acuity. VA was tested in each eye, using the child's current refractive index. The worse-seeing eye was the eye with a lower ETDRS score at the 5th birthday visit. If both eyes had the same ETDRS score, then the left eye was assigned as the worse-seeing eye.
Time Frame: at the participant's fifth birthday visit (maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 45 | 42 | 36
Score on a scale | 60.2 (2.95) | 53.8 (3.05) | 52.2 (3.30)
Statistical Analysis 1: Comparison: Ranibizumab 0.2 mg vs Laser Therapy; Test type: Superiority; ANOVA — P value not applicable because it's a descriptive analysis; Mean Difference (Net) = 8.0, 95% CI 2-sided [-0.8 to 16.7], Standard Error of Mean 4.42
Statistical Analysis 2: Comparison: Ranibizumab 0.1 mg vs Laser Therapy; Test type: Superiority; ANOVA — P value not applicable because it's a descriptive analysis; Mean Difference (Net) = 1.6, 95% CI 2-sided [-7.3 to 10.5], Standard Error of Mean 4.49
Statistical Analysis 3: Comparison: Ranibizumab 0.2 mg vs Ranibizumab 0.1 mg; Test type: Superiority; ANOVA; Mean Difference (Net) = 6.4, 95% CI 2-sided [-2.0 to 14.8], Standard Error of Mean 4.24

5. Secondary Outcome: Number of Participants With Absence of Active Retinopathy of Prematurity (ROP) at 40 Weeks Post Core Baseline Visit
Description: The absence of active ROP in both eyes is defined by the absence of all of the following features: (1) Vessel dilatation of plus disease in at least 2 quardrants (some persisting tortuosity is allowed), (2) Extra-retina vessels extending from the retina into the vitreous and judged to be a sign of active ROP disease.
Time Frame: at 40 weeks post core baseline visit
Population: Extension Safety Set: defined as the subset of the patients from the Safety Set of the core study who entered the extension study and comprised data from both core and extension studies. Number analyzed represents the number of participants with at least one non-missing value for the specific category and, therefore, it's not the same as the total number of participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 57 | 59 | 47
Participants
  Absence of active ROP at 40 weeks post core baseline visit: number analyzed (Participants) | 55 | 58 | 46
  Absence of active ROP at 40 weeks post core baseline visit | 55 | 58 | 46
  Absence of vessel dilatation: number analyzed (Participants) | 55 | 58 | 46
  Absence of vessel dilatation | 55 | 58 | 46
  Absence of extra-retinal vessels | 57 | 59 | 47

6. Secondary Outcome: Number of Participants With Absence of Active Retinopathy of Prematurity (ROP) at 52 Weeks Post Core Baseline Visit
Description: as for outcome 5
Time Frame: at 52 weeks post core baseline visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 58 | 63 | 50
Participants | 58 | 63 | 49

7. Secondary Outcome: Number of Participants With Absence of All Ocular Structural Abnormalities at or Before 40 Weeks Post Baseline Visit
Description: The absence of all ocular structural abnormalities is defined by the absence of all of the following fundus features in both eyes at or before the given time point: (1) Substantial temporal retinal vessel dragging causing abnormal structural features/macular Ectopia, (2) Retrolental membrane obscuring the view of the posterior pole, (3) Posterior retinal fold involving the macula, (4) Retinal detachment involving the macula
Time Frame: at or before 40 weeks post baseline visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants | 59 | 61 | 47

8. Secondary Outcome: Number of Participants With Absence of All Ocular Structural Abnormalities at or Before the Participant's Fifth Birthday Visit
Description: as for outcome 7
Time Frame: at or before the participant's fifth birthday visit (up to maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants | 59 | 61 | 47

9. Secondary Outcome: Number of Participants With Absence of Individual Ocular Structural Abnormalities at or Before 40 Weeks Post Baseline Visit
Description: Number of participants with absence of each structural abnormality in both eyes at or before the given time point: (1) Substantial temporal retinal vessel dragging causing abnormal structural features/macular Ectopia, (2) Retrolental membrane obscuring the view of the posterior pole, (3) Posterior retinal fold involving the macula, (4) Retinal detachment involving the macula, (5) Retinal detachment not involving the macula, (6) Pre-retinal fibrosis
Time Frame: at or before 40 weeks post baseline visit
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants
  Absence of substantial temporal retinal vessel | 59 | 63 | 49
  Absence of Retrolental membrane obscuring the view of the posterior pole | 60 | 65 | 53
  Absence of posterior retinal fold involving the macula | 59 | 65 | 51
  Absence of retinal detachment involving the macula | 60 | 63 | 51
  Absence of retinal detachment not involving the macula | 60 | 62 | 50
  Absence of pre-retinal fibrosis | 58 | 60 | 49

10. Secondary Outcome: Number of Participants With Absence of Individual Ocular Structural Abnormalities at or Before the Participant's Fifth Birthday Visit
Description: Number of participants with absence of each structural abnormality in both eyes at or before the given time point: (1) Substantial temporal retinal vessel dragging causing abnormal structural features/macular Ectopia, (2) Retrolental membrane obscuring the view of the posterior pole, (3) Posterior retinal fold involving the macula, (4) Retinal detachment involving the macula, (5) Retinal detachment not involving the macula, (6) Pre-retinal fibrosis, (7) Optic disc pallor, (8) Optic disc swelling, (9) Pigmentary disturbance in the macula, (10) Atrophic changes in the macula
Time Frame: at or before the participant's fifth birthday visit (up to maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants
  Absence of temporal retinal vessel dragging | 59 | 63 | 49
  Absence of Retrolental membrane obscuring the view of the posterior pole | 60 | 65 | 52
  Absence of posterior retinal fold involving the macula | 59 | 65 | 51
  Absence of retinal detachment involving the macula | 60 | 63 | 50
  Absence of retinal detachment not involving the macula | 60 | 62 | 50
  Absence of pre-retinal fibrosis | 58 | 59 | 48
  Absence of optic disc pallor | 60 | 65 | 52
  Absence of optic disc swelling | 60 | 65 | 53
  Absence of pigmentary disturbance in the macula | 60 | 64 | 52
  Absence of atrophic changes in macula | 60 | 65 | 51

11. Secondary Outcome: Number of Participants With Absence of All Ocular Structural Abnormalities at or Before Participant's 2 Years Corrected Age Visit
Description: as for outcome 7
Time Frame: at or before participant's 2 years corrected age visit (up to 2 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants | 59 | 61 | 47

12. Secondary Outcome: Number of Participants With Absence of Individual Ocular Structural Abnormalities at or Before Participant's 2 Years Corrected Age Visit
Description: as for outcome 10
Time Frame: at or before participant's 2 years corrected age visit (up to 2 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 60 | 65 | 53
Participants
  Absence of substantial temporal retinal vessel dragging | 59 | 63 | 49
  Absence of Retrolental membrane obscuring the view of the posterior pole | 60 | 65 | 52
  Absence of posterior retinal fold involving the macula | 59 | 65 | 51
  Absence of retinal detachment involving the macula | 60 | 63 | 50
  Absence of retinal detachment not involving the macula | 60 | 62 | 50
  Absence of pre-retinal fibrosis | 58 | 59 | 48
  Absence of optic disc pallor | 60 | 65 | 53
  Absence of optic disc swelling | 60 | 65 | 53
  Absence of pigmentary disturbance in the macula | 60 | 64 | 52
  Absence of atrophic changes in macula | 60 | 65 | 52

13. Secondary Outcome: Number of Participants With Recurrence of ROP up to 40 Weeks Post Baseline Visit in the Core Study
Description: Recurrence of ROP was defined as ROP receiving any post-baseline intervention after the 1st study treatment in the core study. In the ranibizumab arms, post-baseline interventions were ranibizumab retreatment or switch to laser. In the laser arm, post-baseline interventions were supplementary laser treatments after 11 days post-baseline, or switch to ranibizumab; supplementary laser treatment within 11 days post-baseline was not counted as recurrence.
Time Frame: up to 40 weeks post baseline visit in the core study
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants | 19 | 22 | 11

14. Secondary Outcome: Number of Participants With Recurrence of ROP up to 52 Weeks Post Baseline Visit in the Core Study
Description: Recurrence of ROP was defined as ROP receiving any post-baseline intervention after the 1st study treatment in the core study. In the ranibizumab arms, post-baseline interventions were ranibizumab retreatment or switch to laser. In the laser arm, post-baseline interventions were supplementary laser treatments after 11 days post-baseline, or switch to ranibizumab; supplementary laser treatment within 11 days post-baseline was not counted as recurrence. Beyond Week 40, participants did not receive any study intervention and no new data was collected after 40 weeks post core baseline visit.
Time Frame: up to 52 weeks post baseline visit in the core study
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants | 19 | 22 | 11

15. Secondary Outcome: Number of Ranibizumab Injections Received Per Participant Over the Whole Safety Observation Period
Description: Number of ranibizumab injections received in the treatment of participants with ROP up to and including 40 weeks post baseline visit in the core study were reported.
Time Frame: up to and including 40 weeks post baseline visit in the core study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of injections
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 11
Number of injections | 2.5 (0.96) | 2.5 (1.06) | 2.4 (0.92)

16. Secondary Outcome: Refraction Status: Summary of Participants at Participant's 2 Years Corrected Age
Description: Summary of participants was reported to evaluate the refraction in each eye at the participant's 2 years corrected age
Time Frame: at participant's 2 years corrected age (maximum 2 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 57 | 54 | 47
diopters
  Best eye | -0.697 (2.7032) | -0.713 (2.6100) | -1.793 (4.1570)
  Worst eye | -0.825 (2.6575) | -0.829 (2.8346) | -1.516 (3.5652)

17. Secondary Outcome: Refraction Status: Summary of Participants at the Participant's Fifth Birthday Visit
Description: Summary of participants was reported to evaluate the refraction in each eye at the participant's 2 years' corrected age
Time Frame: at the participant's fifth birthday visit (maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 52 | 55 | 45
diopters
  Best eye | -0.601 (2.8107) | -0.859 (2.7406) | -1.883 (4.4970)
  Worst eye: number analyzed (Participants) | 52 | 54 | 45
  Worst eye | -0.904 (2.8501) | -1.074 (3.0405) | -1.706 (3.5740)

18. Secondary Outcome: Change From Baseline in Weight
Description: Subject´s weight was reported to evaluate the physical development.
Time Frame: Baseline of the core study, at the subject's 2 years' corrected age (maximum 2 years and 4 months post core baseline visit) and at the subjects' fifth birthday (maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
grams
  Year 2: number analyzed (Participants) | 56 | 58 | 46
  Year 2 | 8695.9 (1406.58) | 8461.7 (1375.95) | 8840.6 (1643.80)
  5th Birthday: number analyzed (Participants) | 52 | 54 | 45
  5th Birthday | 14611.9 (3018.65) | 14324.7 (2616.96) | 14689.4 (3300.05)

19. Secondary Outcome: Change From Baseline in Head Circumference
Description: Subject´s head circumference was reported to evaluate the physical development.
Time Frame: Baseline of the core study and at the subject's 2 years' corrected age (maximum 2 years and 4 months post core baseline visit)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 55 | 56 | 44
cm | 16.5 (2.60) | 16.2 (2.78) | 17.2 (2.81)

20. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure
Description: Subject´s Sitting Diastolic Blood Pressure was reported to evaluate the physical development.
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 38 | 33 | 31
mmHg | 16.7 (14.92) | 13.6 (14.10) | 16.5 (12.14)

21. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure
Description: Subject´s Sitting Systolic Blood Pressure was reported to evaluate the physical development.
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 38 | 32 | 31
mmHg | 20.6 (16.13) | 16.2 (15.95) | 17.6 (12.75)

22. Secondary Outcome: Number of Participants With the Summary of Respiratory Function Status
Description: Number of participants with respiratory function status was reported
Time Frame: at the participants' fifth birthday visit (maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants
  Number of participants with Wheezing/whistling status | 6 | 4 | 2
  Number of participants with attacks of wheezing | 47 | 50 | 45
  Number of participants with frequency of sleep disturbance due to wheezing | 47 | 52 | 47
  Number of participants with presence of wheezing limiting child's speech ability | 1 | 0 | 0
  Number of participants with dry cough status at night | 5 | 2 | 1
  Number of participants with presence of smoker at home | 15 | 8 | 4

23. Secondary Outcome: Number of Participants With Hearing Impairment of Any Type
Description: Number of participants with hearing function status was reported
Time Frame: at the participants' fifth birthday visit (maximum 5 years and 4 months post core baseline visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
Participants | 2 | 2 | 4

24. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization (from birth to first hospital discharge home) was reported to evaluate the health status of the subject
Time Frame: From baseline of the core study up to 5 years and 4 months post core baseline visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 61 | 65 | 54
days | 111.1 (62.27) | 116.2 (78.10) | 95.7 (57.07)

25. Secondary Outcome: Weight at the Time of First Hospital Discharge
Description: Weight (gram) at the time of first hospital discharge was reported to evaluate the health status of the subject
Time Frame: From baseline of the core study up to 5 years and 4 months post core baseline visit
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy
Number analyzed (Participants) | 56 | 62 | 51
gram | 2910.9 (1359.34) | 2966.5 (1198.60) | 2658.7 (926.92)

ADVERSE EVENTS:
Time Frame: throughout the study, up to approximately 5 years
Description: Deaths happened after extension baseline are counted. Serious Adverse Events (SAEs) and Non-SAEs that started during core study and were ongoing at extension baseline or started on/after extension baseline are counted.
Groups:
- Total: Total of all the participants
Arm/Group | Ranibizumab 0.2 mg | Ranibizumab 0.1 mg | Laser Therapy | Total
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/65 | 2/54 | 2/180
Serious Adverse Events (participants affected / at risk) | 21/61 | 27/65 | 26/54 | 74/180
Other Adverse Events (participants affected / at risk) | 41/61 | 46/65 | 40/54 | 127/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.2 mg (N=61) | Ranibizumab 0.1 mg (N=65) | Laser Therapy (N=54) | Total (N=180)
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Eye disorder (Eye disorders) | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2 | 0 | 2
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Retinopathy of prematurity (Eye disorders) | 0 | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 6
Developmental delay (General disorders) | 2 | 0 | 0 | 2
Inflammation (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 1 | 2 | 6
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial food poisoning (Infections and infestations) | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 4 | 3 | 0 | 7
Bronchitis (Infections and infestations) | 3 | 3 | 5 | 11
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 1 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 3
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 1
Herpangina (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 1
Leptospirosis (Infections and infestations) | 0 | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 2
Parainfluenzae viral bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 2 | 1 | 4
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4 | 4 | 10
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2 | 0 | 2
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1 | 2 | 4
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 1 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 1 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 3
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Viral tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Oxygen saturation decreased (Investigations) | 1 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 1 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 1
Febrile convulsion (Nervous system disorders) | 2 | 3 | 0 | 5
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1 | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 1
Periventricular leukomalacia (Nervous system disorders) | 0 | 1 | 0 | 1
Quadriparesis (Nervous system disorders) | 0 | 1 | 0 | 1
Perinatal brain damage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Psychomotor retardation (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 6
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.2 mg (N=61) | Ranibizumab 0.1 mg (N=65) | Laser Therapy (N=54) | Total (N=180)
Astigmatism (Eye disorders) | 3 | 2 | 2 | 7
Myopia (Eye disorders) | 6 | 3 | 5 | 14
Strabismus (Eye disorders) | 10 | 12 | 12 | 34
Constipation (Gastrointestinal disorders) | 4 | 8 | 2 | 14
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4 | 5 | 13
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Developmental delay (General disorders) | 5 | 1 | 3 | 9
Pyrexia (General disorders) | 6 | 11 | 10 | 27
Seasonal allergy (Immune system disorders) | 3 | 2 | 1 | 6
Bronchiolitis (Infections and infestations) | 2 | 3 | 0 | 5
Bronchitis (Infections and infestations) | 4 | 4 | 6 | 14
COVID-19 (Infections and infestations) | 1 | 1 | 3 | 5
Conjunctivitis (Infections and infestations) | 2 | 4 | 4 | 10
Ear infection (Infections and infestations) | 4 | 3 | 0 | 7
Exanthema subitum (Infections and infestations) | 3 | 2 | 1 | 6
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 3 | 5
Influenza (Infections and infestations) | 4 | 2 | 1 | 7
Nasopharyngitis (Infections and infestations) | 11 | 11 | 9 | 31
Otitis media (Infections and infestations) | 7 | 2 | 3 | 12
Pharyngitis (Infections and infestations) | 2 | 3 | 5 | 10
Pneumonia (Infections and infestations) | 5 | 1 | 0 | 6
Respiratory tract infection viral (Infections and infestations) | 3 | 4 | 1 | 8
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5 | 11
Viral upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0 | 3
Iron deficiency (Metabolism and nutrition disorders) | 4 | 0 | 4 | 8
Malnutrition (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Febrile convulsion (Nervous system disorders) | 3 | 2 | 3 | 8
Nystagmus (Nervous system disorders) | 1 | 3 | 1 | 5
Seizure (Nervous system disorders) | 3 | 0 | 2 | 5
Autism spectrum disorder (Psychiatric disorders) | 3 | 1 | 1 | 5
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02640664/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT02640664/SAP_001.pdf